CLINICAL TRIAL: NCT03343808
Title: Pain Treatment With Cooled Radiofrequency in Osteoarthritis and Total Knee Arthroplasty: Case Series in Hospital Universitario de Son Espases
Brief Title: Retrospective Study of the Results of Cooled Radiofrequency for Genicular Nerves Neurotomy in 40 Consecutive Patients With Osteoarthritis of the Knee and Painful Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Hospital Son Espases (Other)
Collaborators: José Andrés López Riquelme (Unknown); María del Pilar Sanchís Cortés (Unknown)
Responsible Party: Principal Investigator, Andrés Camprodón Alberca, Orthopedic Surgeon, Hospital Son Espases
Other Study IDs: 1-2017
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Osteoarthritis, Knee
Keywords: Cooled radiofrequency; chronic knee pain; knee arthroplasty; genicular nerve
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Procedure: cooled radiofrequency ablation of genicular nerves — Cooled RF consists of creating an injury in the nerve trough a high frequency flow. Unlike conventional RF, in cooled RF through a closed circuit where intravenous flows, we can create an injury for a longer period of time, at a lower temperature (standard RFA 90º C, cooled RFA 60º C) and within an area 8 times larger. As the lesion is spherical, and larger (about 10-12 mm in diameter), the chances of neurolysis of the nerve increase.

SUMMARY:
Analyze the results of cooled radiofrequency in patients with chronic knee pain after one year of follow- up.

DETAILED DESCRIPTION:
The investigators performed a retrospective case-series reviewed of 40 patients who underwent cooled RF of genicular nerves. The investigators evaluated results of the survey of quality of life (SF36), knee society score (KSS) and the Visual Analogue Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Chronic knee pain (older than 3 months, with no response to physiotherapy, medication or hyaluronic acid infiltration) with a pain intensity according to VAS>7/10
* The radiological criteria were witness of OA with Kellgren-Lawrence index of 2 to 4.
* Painful TKA with no apparent cause and with a radiological image where a proper placement was observed

Exclusion Criteria:

* Infection or lymphangitis of the member
* Acute knee pain
* Corticoids or hyaluronic acid infiltration with a high molecular weight prior to the surgery
* Pregnancy
* Severe neurological or psychiatric disorders
* Patients with pacemakers

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The procedure was performed to 33 patients with OA (two of them with inflammatory causes) and in 7 patients with TKA (four with revised TKA).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-01-08 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2017-05-26 (Actual)

PRIMARY OUTCOMES:
Treatment success was defined as the number of subjects whose knee pain is reduced by ± 50% based on the Visual Analogue Scale (VAS). | one year after the procedure
  The VAS is a 11- point scale (0 points to 10 points), where 0 points equals "no pain" and 10 points equals the "worst pain".

SECONDARY OUTCOMES:
Short Form (36) Health Survey | one year after the procedure
  The SF36 values eight parameters: physical function, social function, physical role, emotional role, mental health, vitality, pain and general health. Zero is the worst conceivable health and 100 the best.
Knee Society Score (KSS) | one year after the procedure
  The KSS consists of two parts. KS measures pain, range of motion, stability and alignment. FS measures the distance able to walk, the difficulty in going up or down stairs and the need for walking aids. The result is rated as excellent (80-100), good (70-79), regular (60-69) and bad (<60).

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Camprodón Alberca, Principal Investigator — Hospital Son Espases

IPD SHARING:
Plan to Share IPD: Undecided